CLINICAL TRIAL: NCT03194191
Title: Pregnancy With Insomnia: a Trial of Acupuncture
Acronym: GAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P150951
Record Dates: First submitted 2017-05-23; First posted 2017-06-21 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Insomnia
Keywords: Insomnia; Pregnancy; Acupuncture; Insomnia severity index; Pittsburgh Sleep Quality Index; Anxiety; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with regular acupuncture needles vs. sham needles. In addition, the sham needles will be placed in areas that do not correspond to any known acupuncture point.
  5 bilateral acupoints or placebo acupoints,
Who Masked: Participant
Masking Description: Single blind (patient blinded to intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular acupuncture needles (Experimental): Real acupuncture procedure The real acupuncture will be performed by means of standard stainless-steel needles (0.30-mm diameter, 30-mm length/Gauge 8 x 1.2"), located bilaterally in 5 real acupoints.
  Interventions: Device: Acupuncture needles
- Sham acupuncture needles (Sham Comparator): Sham acupuncture with a no penetrating sham needle (blunt and telescopic), giving the impression of insertion but without penetrating the skin will be placed bilaterally in 5 false acupoints
  Interventions: Device: Acupuncture needles

INTERVENTIONS:
Device: Acupuncture needles — The patient will be in a semi recumbent position during needle penetration. Duration of needle insertion: 30 minutes

SUMMARY:
Acupuncture is widely used for treatment of insomnia. The research hypothesis is that acupuncture may be more effective than sham acupuncture to treat insomnia during pregnancy.

GAS is a randomized controlled trial with placebo acupuncture using the insomnia severity index (ISI) as the main outcome criterion.

DETAILED DESCRIPTION:
Scientific justification:

- During pregnancy, insomnia occurs mainly in women without a previous history of sleep disorder, and may remain after delivery. Insomnia affects the quality of life. It might be associated with an increase in labor duration and cesarean section rate.

Insomnia tends to worsen during gestation, owing to back pain, an increased need to micturate, and the movement of the fetus. Sleep disorders are often associated with restless legs syndrome.

* To treat insomnia during pregnancy, the Haute Autorité de Santé (HAS) recommends avoiding using psychotropic medications. It also recommends screening for depression or anxiety traits often associated with insomnia. However, in most cases, psychological means alone fail to treat insomnia effectively.
* Based on 11 randomized controlled trials, the odds of improving sleep disorders are 3 times greater with than without acupuncture, but the methodological quality of these trials is considered insufficient to conclude.

Population:

The study focused on pregnant women suffering from insomnia, excluding women with pregnancies complicated by pre-eclampsia, fetal growth anomalies, or threatened premature labor for fear those complications might interact with sleep disorders, as well as women with known psychiatric disorders. We also excluded women with a history of insomnia before pregnancy to focus on insomnia triggered by pregnancy only.

Objectives:

* Primary objective: To assess the effect of a standardized acupuncture protocol vs. placebo on insomnia during pregnancy.
* Secondary objectives: To assess the effect of a standardized acupuncture protocol vs. placebo on (i) the Pittsburgh Sleep Quality Index (PSQI), (ii) anxiety and depression traits, (iii) use of psychotropic medicines and (iv) recreational substances, (v) the incidence of restless legs syndrome, (vi) perinatal outcome .

Study design:

* Study Type: Multicentre, Interventional, randomized, 2 parallel groups
* Endpoint Classification: Efficacy Study
* Intervention Model: Parallel Assignment
* Masking: Single blind (patient blinded to intervention)
* Primary Purpose: Treatment
* One acupuncture session weekly for 4 consecutive weeks

Visits:

* Selection: When a pregnant woman complains from insomnia, the health professional in charge will fill a checklist of inclusion and exclusion criteria, provide the patient with a pre inclusion ISI questionnaire and give the patient an information sheet and a copy of the consent. When a pregnant woman is sent to the acupuncturist for sleep disorders, he or she may proceed to the selection visit.
* Inclusion: The acupuncturist checks for inclusion and exclusion criteria, collects the patient written consent, performs the clinical examination, gives the corresponding self-assessment questionnaires and proceeds to computerized randomization.
* Follow-up: At visits 1 to 4, the acupuncturist performs the treatment, and records side effects if any. Visits are scheduled on a weekly basis.
* End of research: At visit 5 (one week after last acupuncture session), the acupuncturist gives the corresponding self-assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Singleton pregnancy
* Gestational age ≥ 16 weeks + 0 day and ≤ 32 weeks + 6 days
* Insomnia Severity Index ≥ 10
* Insomnia reported to have started during pregnancy and at least 2 weeks before inclusion
* Patient understanding the study
* Informed consent signed
* Social insurance available at inclusion and until the end of pregnancy

Exclusion Criteria:

* Threatened premature labor
* Small fetus for gestational age
* Pre-eclampsia
* Insomnia starting before pregnancy
* Use of psychotropic drugs before pregnancy
* Use of recreational drugs during pregnancy
* Known psychiatric disorder
* Anticoagulant therapy
* Patient reporting insomnia results from chronic or acute pain
* Obstructive sleep apnea (OSA) requiring treatment
* Patient under antidepressant therapy
* Patient under legal guardianship or deprived of freedom

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index (ISI) | Inclusion visit and 5 weeks after the first acupuncture session
  Difference of ISI self-report questionnaire administrated at inclusion visit and 5 weeks after the first acupuncture session

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Inclusion visit and 5 weeks after the first acupuncture session
  Difference of PSQI self-report questionnaire administrated at inclusion visit and 5 weeks after the first acupuncture session
Hospital Anxiety and Depression Scale (HADS) | Inclusion visit and 5 weeks after the first acupuncture session
  Difference of HADS self-report questionnaire administrated at inclusion visit and 5 weeks after the first acupuncture session
Cumulated dose of each psychotropic medicine | Inclusion visit and 5 weeks after the first acupuncture session
  During the study period, the patients will note on a logbook the daily use of any drug.
Cumulated dose of alcohol | Inclusion visit and 5 weeks after the first acupuncture session
  During the study period, the patients will note on a logbook the daily use of alcohol.
Cumulated dose of tobacco | Inclusion visit and 5 weeks after the first acupuncture session
  During the study period, the patients will note on a logbook the daily use of tobacco.
Cumulated dose of cannabis | Inclusion visit and 5 weeks after the first acupuncture session
  During the study period, the patients will note on a logbook the daily use of cannabis.
Cumulated dose of other recreational substances or medicine | Inclusion visit and 5 weeks after the first acupuncture session
  During the study period, the patients will note on a logbook the daily use of other recreational substances and medicine.
Difference in the frequency of restless leg syndrome | Inclusion visit and 5 weeks after the first acupuncture session
  According to the guidelines of the International Restless Legs Syndrome Study Group.
  The diagnosis of restless leg will rely on the presence of all of the following criteria:
  1. Desire to move the extremities usually associated with discomfort or disagreeable sensations in the extremities.
  2. Motor Restlessness-patients move to relieve the discomfort, for example walking, or to provide a counter-stimulus to relieve the discomfort, for example, rubbing the legs.
  3. Symptoms are worse at rest with at least temporary relief by activity.
  4. Symptoms are worse later in the day or at night.
Perinatal outcome - Gestational age at birth | At birth
  The gestational age at birth of the newborn will be recorded.
Perinatal outcome - birth weight | At birth
  The weight (in gr) at birth of the newborn will be recorded.
Perinatal outcome - birth height | At birth
  The height (in cm) at birth of the newborn will be recorded.
Perinatal outcome - sex | At birth
  The sex of the newborn will be recorded.
Perinatal outcome - perinatal mortality | At birth
  The perinatal mortality will be recorded.
Perinatal outcome - five minutes Apgar score | At birth
  The five minutes Apgar score will be recorded.
Perinatal outcome - cesarean section rate | At birth.
  Cesarean section rate will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Nicolian, Midewife, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No